CLINICAL TRIAL: NCT04044222
Title: A Phase III, Multicenter, Randomized, Double-Blind, Placebo-Controlled Trial Comparing the Efficacy and Safety of a Sintilimab Plus ICE Regimen Versus a Placebo Plus ICE Regimen in Classic Hodgkin's Lymphoma Patients With First-line Standard Chemotherapy Failure
Brief Title: A Study to Evaluate the Efficacy and Safety of a Sintilimab Plus ICE Regimen Versus ICE Regimen in Classic Hodgkin's Lymphoma Patients (cHL) Who Have Failed First-line Standard Chemotherapy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CIBI308B301
Record Dates: First submitted 2019-08-01; First posted 2019-08-05 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Classic Hodgkin's Lymphoma
MeSH Terms: interventions — sintilimab; Carboplatin; Etoposide; Ifosfamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Sintilimab, etoposide, ifosfamide, carboplatin) (Experimental): Patients receive sintilimab IV on day 1, etoposide IV on days 1-3 of courses 1-6, carboplatin IV on day 2 of courses 1-6, and ifosfamide IV on day 1-3 of courses 1-6. Sintilimab in combination with ICE chemotherapy repeats every 21 days for 6 courses.
  Interventions: Biological: Sintilimab; Drug: Carboplatin; Drug: Etoposide; Drug: Ifosfamide
- Treatment (placebo, etoposide, ifosfamide, carboplatin) (Experimental): Patients receive placebo IV on day 1, etoposide IV on days 1-3 of courses 1-6, carboplatin IV on day 2 of courses 1-6, and ifosfamide IV on day 1-3 of courses 1-6. Placebo in combination with ICE chemotherapy repeats every 21 days for 6 courses.
  Interventions: Drug: Placebo; Drug: Carboplatin; Drug: Etoposide; Drug: Ifosfamide

INTERVENTIONS:
Biological: Sintilimab — IV
  Arms: Treatment (Sintilimab, etoposide, ifosfamide, carboplatin)
Drug: Carboplatin — IV
  Arms: Treatment (Sintilimab, etoposide, ifosfamide, carboplatin)
Drug: Etoposide — IV
  Arms: Treatment (Sintilimab, etoposide, ifosfamide, carboplatin)
Drug: Ifosfamide — IV
  Arms: Treatment (Sintilimab, etoposide, ifosfamide, carboplatin)
Drug: Placebo — IV
  Arms: Treatment (placebo, etoposide, ifosfamide, carboplatin)
Drug: Carboplatin — IV
  Arms: Treatment (placebo, etoposide, ifosfamide, carboplatin)
Drug: Etoposide — IV
  Arms: Treatment (placebo, etoposide, ifosfamide, carboplatin)
Drug: Ifosfamide — IV
  Arms: Treatment (placebo, etoposide, ifosfamide, carboplatin)

SUMMARY:
This phase III trial studies the side effects of sintilimab to see how well it works when given together with ifosfamide, carboplatin, and etoposide in treating patients with classic Hodgkin lymphoma that does not respond to first-line standard chemotherapy.

DETAILED DESCRIPTION:
randomized, double-blind, two arms , multicenter

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Histopathologically confirmed cHL
3. Failed first-line standard combination chemotherapy
4. One measurable lesion (Lugano 2014)
5. Eastern Cooperative Oncology Group (ECOG) of 0-1
6. Male or female aged ≥18 years
7. Patients must have adequate organ and bone marrow function

Exclusion Criteria:

1. Patients must not have known central nervous system (CNS) involvement
2. Patients must not have had prior exposure to any immune checkpoint inhibitors including anti-PD-L1 agents, anti-PD-L2 agents, or anti-CTLA-4 monoclonal antibodies
3. Patients may not simultaneously participate in another interventional clinical study
4. Patients may not receive any other investigational agents within 4 weeks of study registration
5. Patients may not receive any other form of immunosuppressive therapy within 4 weeks prior to the first dose of study drug
6. Patients may not receive live attenuated vaccines within 4 weeks prior to the first dose of study drug (or plan to receive live attenuated vaccines during the study period)
7. Patients with known immunodeficiency are ineligible
8. Patients with known active TB (Bacillus tuberculosis) are ineligible
9. Patients must not have had prior allogeneic stem cell transplantation or allogeneic organ transplantation
10. Patients must not be pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2019-10-21 (Actual); Primary Completion 2023-07-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
PFS | 44months

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China